CLINICAL TRIAL: NCT04034784
Title: Controlled, Single Ascending Volume Clinical Trial to Evaluate the Safety and Tolerability of the Adhesion Reduction Medical Device Discrete(TM) in Healthy Volunteers
Brief Title: Discrete(TM) Safety Clinical Trial GLAD-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARC Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ARCMD-GLAD-01; GLAD-01 (Other: ARC Medical Devices Inc.)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Safety and Tolerability in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discrete(TM) (Experimental): Intraperitoneal injection
  Interventions: Device: Discrete(TM)
- Control Lactated Ringer's Solution (Control LRS) (Sham Comparator): Intraperitoneal injection
  Interventions: Other: Control Lactated Ringer's Solution (Control LRS)

INTERVENTIONS:
Device: Discrete(TM) — A designated volume of Discrete(TM) (according to cohort) is applied intraperitoneally
  Arms: Discrete(TM)
Other: Control Lactated Ringer's Solution (Control LRS) — A designated volume of LRS (according to cohort and equivalent to volume of Discrete(TM)) is applied intraperitoneally
  Arms: Control Lactated Ringer's Solution (Control LRS)

SUMMARY:
This study will assess the safety and tolerability of a new liquid anti-adhesion device, Discrete(TM), in healthy volunteers, in order to determine the best volume of Discrete(TM) to go forward into clinical efficacy research.

The clinical trial will progress in accordance with first-in-human study guidance from the United States Food and Drug Administration (US FDA) and European Medicines Agency (EMA).

It will be conducted as a randomized, controlled, double-blinded, single ascending volume, single-center, interventional safety trial. Participants will remain blinded to treatment until end of clinical trial. A maximum of 7 cohorts will be studied to assess maximum tolerated volume of investigational medical device compared with Control Lactated Ringer's solution (LRS) administered intraperitoneally. The trial will commence with a low volume and progress in a sequential, stepwise volume-escalating schema until defined maximum tolerated volume criteria are met. Following determination of the maximum tolerated volume, it is anticipated that up to 2 additional cohorts will be enrolled, wherein all participants will also receive a single standard dose of a commonly used anticoagulant as used in surgeries.

A maximum of 81 participants will be enrolled. Eligible and consented adult men and women will be sequentially enrolled within each cohort at a ratio of 6 participants on Discrete(TM) to 3 participants on Control LRS. Participants will be followed for up to 10 days after intraperitoneal application.

An independent Data and Safety Monitoring Committee will closely review safety in the clinical trial.

ELIGIBILITY:
Pre-Application Inclusion criteria

* Understand and be able to follow the requirements of the protocol including signing and dating an REB approved Informed Consent Form prior to undergoing any protocol related procedures
* Adult healthy volunteers ≥ 18 to ≤ 60 years of age, male or female

  * Female participants must fulfil one (1) of the following criteria:

    i) Post-menopausal; defined as either amenorrhea ≥ 12 months and confirmed with follicle stimulating hormone test ii) Females of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from at least 30 days before the study and for the duration of the study until 45 days post-intraperitoneal treatment. Adequate contraception includes:
    1. hormonal implant combined with a barrier method (male or female condom diaphragm with spermicidal foam/gel/film/cream/suppository or cervical cap with spermicide).
    2. intrauterine system (IUS) combined with a barrier method (male or female condom diaphragm with spermicidal foam/gel/film/cream/ suppository or cervical cap with spermicide).
    3. intrauterine device (IUD) combined with a barrier method (male or female condom diaphragm with spermicidal foam/gel/film/cream/ suppository or cervical cap with spermicide).
    4. hormonal patch combined with a barrier method (male or female condom diaphragm with spermicidal foam/gel/film/cream/ suppository or cervical cap with spermicide).
    5. hormonal contraceptive pills combined with a barrier method (male or female condom diaphragm with spermicidal foam/gel/film/cream/ suppository or cervical cap with spermicide).
    6. double-barrier methods (e.g., male condom with diaphragm and spermicide, male condom with cervical cap and spermicide).
    7. complete abstinence as a method of contraception is acceptable if in line with the subject's usual and preferred lifestyle.
  * Male subjects who are non-vasectomized (or vasectomized less than six (6) months prior device application) and have female partners of childbearing potential must be willing to tell their female partner(s) that they are participating in a research study, and use an effective birth control method when having heterosexual intercourse, from treatment application until 45 days post-intraperitoneal treatment. Effective methods of contraception for use by males include:

    i) using a condom with a female partner of child-bearing potential who is using oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicidal foam/gel/film/ cream/suppository.

ii) complete abstinence as a method of contraception is acceptable if in line with the subject's usual and preferred lifestyle.

* In good general health as evaluated by the Principal Investigator
* Has undergone a satisfactory physical and medical assessment with no clinically significant and relevant abnormalities, comorbidities, chronic or acute infections
* No history of previous abdominopelvic surgery including laparoscopy, laparotomy, caesarean section, or other access that could have resulted in development of adhesions
* No symptoms, history, treatment or prior diagnosis of endometriosis, pelvic inflammatory disease, chlamydia, polycystic ovaries, inflammatory bowel disease, diverticulitis, irritable bowel syndrome or other condition likely to result in abdominopelvic inflammation or sensitivity, or development of adhesions
* Have a negative pregnancy test within 1 day (24 hours) of device or control application (female participants only)
* Is willing, able and likely to fully comply with clinical trial procedures and restrictions including follow-ups

Pre-Application Exclusion Criteria

* Are unable to give their own written informed consent
* Current pregnancy including ectopic pregnancy within last 6 months (including any previous ectopic pregnancy treated surgically) (female participants only)
* Positive pregnancy test (female participants only)
* Are breastfeeding (female participants only)
* Are within 3 months post-partum (female participants only)
* Are anticipated to attempt pregnancy within 45 days after intraperitoneal application
* Participant has donated blood in the following volumes:

  i) Between 50 mL and 499 mL within 30 days prior to the screening visit ii) 500 mL or more within 60 days prior to the screening visit
* Participant has a BMI of ≤ 18.5 or ≥ 30, and in the opinion of the Investigator does not have - Has undergone previous abdominopelvic surgery including laparoscopy, laparotomy, caesarean section, or other access that could have resulted in development of adhesions
* Has had symptoms, history, treatment or prior diagnosis of any inflammatory condition affecting the abdominopelvic cavity, including; endometriosis, pelvic inflammatory disease, chlamydia, polycystic ovaries, inflammatory bowel disease (including Crohn's disease, Ulcerative Colitis and Microscopic colitis), diverticulitis, irritable bowel syndrome, intestinal obstructive disease or other condition likely to result in abdominopelvic inflammation or sensitivity, or development of adhesions
* Have diabetes
* Have clinically significant abnormal blood results as reviewed by Principal Investigator
* Have creatinine clearance <30 mL/min as per Cockcroft-Gault equation
* Concurrent use or anticipated use of systemic corticosteroids, antineoplastic agents within 2 months of intraperitoneal application
* Participant has received immunosuppressant therapy within last 30 days
* Have had previous radiation therapy in thoracic or abdominopelvic cavity
* History of malignancy (excluding basal cell carcinoma)
* History of heparin-induced thrombocytopenia (HIT) or known sensitivity to heparin-like products (including enoxaparin sodium)
* Have clinically relevant hemochromatosis, hepatic, renal, autoimmune, lymphatic, - Family history of blood or coagulation disorders
* Have any concomitant medical treatment including anticoagulant therapy, over-the-counter medications and/or herbal supplements or teas within preceding 14 days of clinical trial unit - Active pelvic or abdominal infection or other active infection with fever greater than 37.6°C
* Known or suspected allergy to brown seaweed, food allergies and/or presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant"
* Any other severe allergic conditions (e.g., anaphylactic reactions, angioedema)
* Currently enrolled in another clinical study/trial or has been in another study within the last 30 days
* Have received or is expected to receive any investigational product or investigational technique within 30 days prior to or during enrolment
* Participants who are, in the opinion of the Investigator, unable to comply with the clinical trial schedule and protocol evaluations
* Participants who, in the opinion of the Investigator, would not be suitable for clinical trial participation
* Participants with clinically significant ECG or other screening visit abnormality that, in the opinion of the Investigator, would not be suitable for clinical trial participation
* Participant has current or any history of prior bladder or urinary injury; or history of recurrent bladder or urinary problems, including recurrent urinary tract infections in last 12 months; or a single occasion bladder or urinary problem, including cystitis or proven urinary tract infection within the last 3 months
* Participant has suspected abdominal abscess
* Have a positive methicillin-resistant Staphylococcus aureus (MRSA) test at screening only
* A known history or positive test result for human immunodeficiency virus (HIV), chronic Hepatitis B surface antigen, or Hepatitis C antibody at screening only.
* Evidence of alcohol or substance abuse, or previous alcohol or substance abuse
* Participant not willing to refrain from use of alcohol throughout clincial trial unit admission and for 48 hours prior to any clinic visit.
* A positive urine drug screen (Marijuana, Amphetamines, Phencyclidine, Barbiturates, Cocaine, Opiates, Benzodiazepines).
* Participant not willing to refrain from egg donation from time of consent to 45 days after
* Participant not willing to refrain from sperm donation from time of consent to 45 days after intraperitoneal application (male participants only)
* Participant not willing to refrain from smoking or using any tobacco/nicotine-containing products from at least 6 months prior to study device application and for the entire duration of the study.
* Participant not willing to refrain from strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) for at least 72 hours prior to admission to the
* Participant has a history of or has a current hernia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Safety as evaluated by assessment of adverse events in treatment and control group | Up to 10 days post application
  The rate of adverse events will be compared in treatment and control groups

SECONDARY OUTCOMES:
Participant recovery | Post application to 10 days post application
  Participant recovery after Discrete(TM) application

CONTACTS AND LOCATIONS:
Overall Officials: Chris Springate, PhD, Study Director — ARC Medical Inc.
Locations (1):
- Clinical trial site, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No